CLINICAL TRIAL: NCT02139098
Title: Phase III Study on Alternative Dosing Regimens in the Pharmacotherapy of Mild to Moderate Insomnia
Brief Title: Alternative Dosing Regimens in the Pharmacotherapy of Insomnia
Acronym: ALPHASOM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruiting problems because of the time expenditure required for participating and the strict criteria of inclusion and exclusion
Sponsor: Philipps University Marburg (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Philipps University Marburg Coordination Centre for Clinical Trials (Unknown)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOR1328-SP8; 2013-003229-27 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-05-15 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Insomnia
Keywords: sleep architecture; conditioning of pharmacological responses; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Amitriptyline; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Amitriptyline flexible dosing (Experimental): 50 mg capsule amitriptyline before going to bed on 8 out of 17 nights/placebo
  Interventions: Drug: Amitriptyline; Drug: Placebo
- Zolpidem flexible dosing (Experimental): 5 mg capsule zolpidem before going to bed on 8 out of 17 nights/placebo
  Interventions: Drug: Zolpidem; Drug: Placebo
- Amitriptyline fixed dosing (Active Comparator): 50 mg capsule amitriptyline before going to bed on 8 out of 17 nights
  Interventions: Drug: Amitriptyline
- Zolpidem fixed dosing (Active Comparator): 5 mg capsule zolpidem before going to bed on 8 out of 17 nights
  Interventions: Drug: Zolpidem
- Amitriptyline continuous dosing (Active Comparator): 50 mg capsule amitriptyline before going to bed on 13 out of 17 nights
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline — 50 mg capsule amitriptyline before going to bed on 8 out of 17 nights
  Arms: Amitriptyline fixed dosing; Amitriptyline flexible dosing
Drug: Zolpidem — 5 mg capsule zolpidem before going to bed on 8 out of 17 nights
  Arms: Zolpidem fixed dosing; Zolpidem flexible dosing
Drug: Amitriptyline — 50 mg capsule amitriptyline before going to bed on 13 out of 17 nights
  Arms: Amitriptyline continuous dosing
Drug: Placebo — Placebo
  Arms: Amitriptyline flexible dosing; Zolpidem flexible dosing

SUMMARY:
The purpose of this study is to evaluate whether drug efficiency of zolpidem and amitriptyline can be conditioned according to learning theory in patients with primary insomnia.

DETAILED DESCRIPTION:
Previous research has shown that repeated drug treatments can be regarded as conditioning processes. Sleep disorders are especially of interest to be investigated under the perspective of conditioning with drugs, since sleep quality can be defined both in terms of subjective ratings (self-rated sleep quality parameters) and objective measures (via polysomnographic assessment PSG; e.g., total sleep time, sleep onset, sleep architecture). By using two different drugs (zolpidem, amitriptyline) that modulate sleep differentially, the investigators intend to implement a conditioning paradigm in sleep disorders dissociating conditioning effects on subjective and objective sleep parameters. Both drugs should affect objective and subjective sleep parameters positively, while only amitriptyline should modulate the objectively assessed sleep architecture by REM-suppression (latency of REM-sleep onset, percentage of REM-sleep).Patients with mild to moderate insomnia will undergo a classical conditioning paradigm with one of two study medications: amitriptyline or zolpidem. After an acquisition period and a wash-out period, conditioned sleep changes are assessed in an evocation trial. During a second treatment phase of 7 days, patients receive different doses of amitriptyline (between 0mg and 50mg per night) or zolpidem (between 0mg and 5mg per night) to evaluate alternative dosing regimens in the pharmacotherapy of mild to moderate Insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 years to 69 years
2. fluent in German language
3. provide written informed consent
4. ability to understand the explanations and instructions given by the study physician and the investigator

Exclusion Criteria:

1. Sleep disorders caused by medical factors (e.g. sleep apnea, restless legs syndrome, narcolepsy, substance-induced insomnia)
2. Contraindications to study medication intake according to the information sheet for health professionals (Summary of medicinal Product Characteristics, SmPC; Fachinformation in Germany) assessed by physical examination (including ECG) and medical history

   * allergies to amitriptyline hydrochloride or any of its ingredients
   * allergies to zolpidem or any of its ingredients
   * acute intoxication with alcohol, analgetics, hypnotics or any other psychotropic drug
   * urinary retention
   * delirium
   * untreated closed-angle glaucoma
   * prostatic hyperplasia
   * pyloric stenosis
   * paralytic ilius
   * suicidal thoughts
   * liver/ kidney/ pulmonary insufficiency
   * myasthenia gravis
   * hypokalemia
   * bradycardia
   * coronary heart disease, cardiac arrhythmias, long QT syndrome or other clinically relevant cardiac disorders
   * increased risk of seizures/ history of seizures
   * substance dependence syndrome/ history of substance dependence syndrome
3. Allergies to ingredients of placebo or novel-tasting drink (CS)
4. currently pregnant (verified by urine pregnancy test) or lactating
5. patients scoring ≥12 on the Epworth Sleepiness Scale
6. patients scoring below 8 or above 21 on the Insomnia Severity Index
7. patients suffering from a mental disorder as verified by the SCID (major depression; psychosis; brain injury; substance abuse or dependency syndrome during the last 6 months before V1)
8. nicotine consumption > 10 cigarettes/day
9. unwillingness to refrain from alcohol consumption throughout the study
10. Concomitant medication interfering with study medication intake due to potential interactions (all psychotropic medication including analgetics and muscle relaxants, hypericum derivatives; antihypertensives; anti-arrhythmic agents; antibiotics; cisaprid; anti-malaria drugs; diuretics; imidazole antifungals; cumarin derivatives; antihistaminics; calcium channel blockers; medications that enlarge the QT interval or may lead to hypokalemia)
11. change in concomitant medication regime during the last 2 weeks prior to visit 1 or after randomization
12. intake of psychotropic medication during the last 3 months
13. participation in any other clinical trial 3 months prior to visit 1
14. women of childbearing age not using 2 highly effective contraceptive methods
15. employee of the Sponsor or the principal investigator

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Objective Total Sleep Time | Change from baseline to day 10 after first medication intake
  assessed by polysomnography
Objective Sleep Onset Latency | Change from baseline to day 10 after first medication intake
  assessed by polysomnography
Self-reported Total Sleep Time | Change from baseline to day 10 after first medication intake
  assessed by sleep diary
Self-Reported Sleep Onset Latency | Change from baseline to day 10 after first medication intake
  assessed by sleep diary

SECONDARY OUTCOMES:
Percentage of REM sleep | Change from baseline to day 10 after first medication intake
  assessed by polysomnography
REM onset latency | Change from baseline to day 10 after first medication intake
  assessed by polysomnography
Objective Sleep Efficiency | Change from baseline to day 17 after first medication intake
  assessed by actigraphy
Objective Total Sleep Time | Change from baseline to day 17 after first medication intake
  assessed by actigraphy
Self-Reported Total Sleep Time | Change from baseline to day 18 after first medication intake
  assessed by sleep diary
Self-reported Sleep Onset Latency (min) | Change from baseline to day 18 after first medication intake
  assessed by sleep diary
Self-reported Sleep Onset Latency (evaluation) | Change from baseline to day 18 after first medication intake
  assessed by sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Clinical Psychology and Psychotherapy, Department of Psychology, Philipps University Marburg; Bettina K Doering, Dr., Principal Investigator — Clinical Psychology and Psychotherapy, Department of Psychology, Philipps University Marburg; Carmen Schade-Brittinger, Study Chair — Koordinierungszentrum für Klinische Studien Marburg, Philipps University Marburg
Locations (1):
- Clinical Psychology and Psychotherapy, Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany